CLINICAL TRIAL: NCT05571761
Title: Feasibility and Usefulness of a Neuropsychological Telerehabilitation Program in Asymptomatic HIV Patients: Pilot Randomized Controlled Trial
Brief Title: Teleneuropsychological Intervention in Asymptomatic HIV Seropositive Patients: N&C NeuroChange
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: experimental abandonment
Sponsor: Universidad Nacional Autonoma de Mexico (Other)
Responsible Party: Principal Investigator, Natalia Cortés Corona, MD, Principal Investigator, Universidad Nacional Autonoma de Mexico
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TNSP
Record Dates: First submitted 2022-09-27; First posted 2022-10-07 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Telerehabilitation; Neuropsychology; HIV Dementia
Keywords: HIV; HAND; Teleneuropsychological intervention
MeSH Terms: conditions — AIDS Dementia Complex

STUDY DESIGN:
Intervention Model Description: A pilot randomized clinical trial will be conducted with HIV+ participants randomised in a 1:1 ratio to a study group that will receive the neuropsychological intervention and a second control group that will remain waiting until the study group finishes the intervention and after that can receive the intervention.
Who Masked: Participant
Masking Description: Random assignment will not be disclosed to the participants. The participants in the intervention arm will be contacted first, and once this is completed, the participants in the waiting list control arm will be contacted for the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Refers to the experimental group that will receive the cognitive stimulation program intervention.
  Interventions: Behavioral: Cognitive stimulation program
- Waiting list control group (Other): Will be the control group that remains without intervention until the study group completes the cognitive stimulation program and the subsequent neuropsychological assessment has been done. Once the intervention is completed with the study group, the same program will be applied to the control group.
  Interventions: Behavioral: Cognitive stimulation program

INTERVENTIONS:
Behavioral: Cognitive stimulation program — The cognitive stimulation program consists of 12 sessions of approximately 45 minutes, distributed in a first stage of training and psychoeducation (1 session), a second stage to address emotional aspects of anxiety and depression (2 sessions), and neuropsychological training (8 sessions) and a final closing stage with one session. There will be two sessions per week for 6 weeks.
  The neuropsychological training includes 20 activities whose level of difficulty will vary according to the number of stimuli and the time of stimuli presentation. It includes 5 attentional activities, 3 memory activities, 5 executive functioning activities, one visuospatial skills activity and 6 ecological activities. These activities will be developed on a digital computer platform where patients will be assigned an identification and password to ensure confidentiality.
  Other Names: N&C NeuroChange

SUMMARY:
Currently 37.9 million people are living with human immunodeficiency virus (HIV) around the world (UNAIDS, 2018). Even with antiretroviral treatment (ART), the virus enters the central nervous system and can affect the following structures: amygdala, hippocampus, thalamus, parietal, frontal, temporal regions, orbitofrontal, cingulate, motor and sensory cortex; generating cognitive, behavioral and motor alterations, up to HIV-associated neurocognitive disorder (HAND) and occasionally HIV-associated dementia (HAD).

Few clinical studies have been conducted using computerized cognitive rehabilitation programs to counteract neuropsychological alterations. The aim of this project is to explore the feasibility of a cognitive stimulation program (CSP) developed to strengthen cognitive domains identified as impaired through a neuropsychological assessment in asymptomatic HIV+ patients adherent to ART, with the purpose of improving their quality of life and mood disorder.

DETAILED DESCRIPTION:
A pilot randomized controlled trial (RCT) will be conducted with a study group and a control group in waiting list. This design will be used because it allows to evaluate the feasibility of a teleneuropsychological intervention (N&C NeuroChange) and to identify a preliminary effect as a first approach in a given population, provides greater experimental control over the study variables and allows pre-intervention, post-intervention and follow-up comparisons.

Lancaster et al. (2004) state that n=30 is acceptable for a pilot study, while (Julious, 2005) suggest a minimum sample of n=12 per group. Therefore, 24 participants will be recruited for this study. This has already been implemented in other pilot studies that sought to identify the efficacy of an intervention using samples of 20 (Berrymam et al., 2020) and 13 participants (Delaney, 2018) in total. Although the size of the sample may be a methodological limitation, it will be considered in the discussion of the results; in addition to being a preliminary study to carry out a more rigorous study with an RCT. Participants will be eligible if they are between 20 and 45 years old because 77.5% of the reported cases are in this age range in Mexico (CENSIDA, 2022) .

The procedure will be as follows: All participants will be explained what the study consists of, the intervention and will be given informed consent. Patients will be recruited from the Specialized Clinic Condesa Iztapalapa that serves people living with HIV. A brief medical history will begin with an interview to collect medical history (HIV pathological and infectious history such as time of evolution, viral load, CD4 level, ART regimen, as well as substance abuse and cognitive complaints) and then a neuropsychological assessment will be performed. With those candidates who meet the inclusion criteria and wish to participate, will be randomly assigned in a 1:1 ratio to the intervention group or waiting list control arm. The intervention will begin first with the study group, and a subsequent evaluation will be carried out and then the intervention will be applied to the control group on the waiting list, which will also undergo a subsequent evaluation. Both groups will undergo a third follow-up evaluation three months later to identify whether the changes were maintained over time. Main outcomes of interest include evaluation of the achievement of intervention objectives, usability and acceptability of the CSP. Baseline and follow up measures include assessment of attention, memory, visuospatial skills, working memory, processing speed, verbal fluency, planning, abstraction, depressive and anxiety symptomatology, and daily functionality.

ELIGIBILITY:
Inclusion Criteria:

* Male or females with HIV
* Minimum primary education
* From 20 to 45 years old
* Normal or corrected vision and hearing
* Treatment adherence

Exclusion Criteria:

* Neurological and psychiatric history (except mood disorders)
* Head injuries
* Cerebrovascular events
* Substance abuse
* AIDS associated diseases
* Hormonal therapy

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Attention | Baseline
  Direct digits of the Integrated Neuropsychological Exploration Program. The repetition of a series of digits is requested and an element is added as the task progresses. Uses percentile scores.
Memory | Baseline
  Immediate and deferred texts, and word learning of the Integrated Neuropsychological Exploration Program. Two stories are read and at the end of each one, the patient is asked to narrate everything he/she remembers from the story. In case of not remembering elements, questions are asked about the missing information. The stories are asked again after 5 minutes. Uses percentile scores.
Visuospatial skills | Baseline
  Rey Figure of the NEUROPSI A&M. A complex figure is copied from a model. Afterwards, the figure is drawn again without the model. Uses scalar scores.
Working memory | Baseline
  Digits and letters of the Weschler Adults Intelligence Scale IV. Numbers and letters are provided in disorder and all the elements are asked to be repeated in order, first the numbers and then the letters. Uses scalar scores.
Processing speed | Baseline
  Word reading of Stroop test. A list of 5 columns of words with 20 items each is read as quickly as possible. Uses percentile scores.
Verbal fluency | Baseline
  Categorical recall of the Integrated Neuropsychological Exploration Program. The highest number of animals is said in one minute and the highest number of words beginning with "p" in three minutes. Uses percentile scores.
Planning | Baseline
  Zoo test of the Behavioral Assessment of Dysexecutive Syndrome and Behavioral Rating Inventory of Executive Functioning for Adults. Consists in marking a route in a zoo map to visit different places. Afterwards, the person marks again in the zoo map a rout but is told which route to follow.
Abstraction | Baseline
  Resemblances of the Weschler Adults Intelligence Scale IV. Consists in mentioning what two words have in common or how they are similar. Uses scalar scores.
Attention | Immediately after the intervention
  Direct digits of the Integrated Neuropsychological Exploration Program. The repetition of a series of digits is requested and an element is added as the task progresses. Uses percentile scores.
Memory | Immediately after the intervention
  Immediate and deferred texts, and word learning of the Integrated Neuropsychological Exploration Program. Two stories are read and at the end of each one, the patient is asked to narrate everything he/she remembers from the story. In case of not remembering elements, questions are asked about the missing information. The stories are asked again after 5 minutes. Uses percentile scores.
Visuospatial skills | Immediately after the intervention
  Rey Figure of the NEUROPSI A&M. A complex figure is copied from a model. Afterwards, the figure is drawn again without the model. Uses scalar scores.
Working memory | Immediately after the intervention
  Digits and letters of the Weschler Adults Intelligence Scale IV. Numbers and letters are provided in disorder and all the elements are asked to be repeated in order, first the numbers and then the letters. Uses scalar scores.
Processing speed | Immediately after the intervention
  Word reading of Stroop test. A list of 5 columns of words with 20 items each is read as quickly as possible. Uses percentile scores.
Verbal fluency | Immediately after the intervention
  Categorical recall of the Integrated Neuropsychological Exploration Program. The highest number of animals is said in one minute and the highest number of words beginning with "p" in three minutes. Uses percentile scores.
Planning | Immediately after the intervention
  Zoo test of the Behavioral Assessment of Dysexecutive Syndrome and Behavioral Rating Inventory of Executive Functioning for Adults. Consists in marking a route in a zoo map to visit different places. Afterwards, the person marks again in the zoo map a rout but is told which route to follow.
Abstraction | Immediately after the intervention
  Resemblances of the Weschler Adults Intelligence Scale IV. Consists in mentioning what two words have in common or how they are similar. Uses scalar scores.
Attention | Up to 12 weeks
  Direct digits of the Integrated Neuropsychological Exploration Program. The repetition of a series of digits is requested and an element is added as the task progresses. Uses percentile scores.
Memory | Up to 12 weeks
  Immediate and deferred texts, and word learning of the Integrated Neuropsychological Exploration Program. Two stories are read and at the end of each one, the patient is asked to narrate everything he/she remembers from the story. In case of not remembering elements, questions are asked about the missing information. The stories are asked again after 5 minutes. Uses percentile scores.
Visuospatial skills | Up to 12 weeks
  Rey Figure of the NEUROPSI A&M. A complex figure is copied from a model. Afterwards, the figure is drawn again without the model. Uses scalar scores.
Working memory | Up to 12 weeks
  Digits and letters of the Weschler Adults Intelligence Scale IV. Numbers and letters are provided in disorder and all the elements are asked to be repeated in order, first the numbers and then the letters. Uses scalar scores.
Processing speed | Up to 12 weeks
  Word reading of Stroop test. A list of 5 columns of words with 20 items each is read as quickly as possible. Uses percentile scores.
Verbal fluency | Up to 12 weeks
  Categorical recall of the Integrated Neuropsychological Exploration Program. The highest number of animals is said in one minute and the highest number of words beginning with "p" in three minutes. Uses percentile scores.
Planning | Up to 12 weeks
  Zoo test of the Behavioral Assessment of Dysexecutive Syndrome and Behavioral Rating Inventory of Executive Functioning for Adults. Consists in marking a route in a zoo map to visit different places. Afterwards, the person marks again in the zoo map a rout but is told which route to follow.
Abstraction | Up to 12 weeks
  Resemblances of the Weschler Adults Intelligence Scale IV. Consists in mentioning what two words have in common or how they are similar. Uses scalar scores.

SECONDARY OUTCOMES:
Depressive Symptoms | Baseline
  Patient Health Questionnaire - 9. A self-applied questionnaire that identifies the presence of depressive symptomatology based on a Likert-type scale of 9 items. Based on the cut-off points, minimal (0-4), mild (5-9), moderate (10-14), moderate to severe (15-19) and severe (20-27) depression can be identified.
Anxiety symptoms | Baseline
  General Anxiety Disorder - 7. A self-applied scale to identify generalized anxiety. It consists of a self-applied questionnaire of seven Likert-type questions. Based on the cut-off points, no anxiety (0-4), mild anxiety symptoms (5-9), moderate anxiety symptoms (10-14) and severe anxiety symptoms (15-21) can be identified.
Daily functionality | Baseline
  The Activities of Daily Living Questionnaire. This instrument evaluates daily functioning by assessing basic and instrumental activities in six areas (self-care, home activities, work, recreation, money management, travel and communication, and information technology); it is usually useful for patients with mild cognitive or motor limitations. It allows to generate a percentage of functional impairment by adding the scores of each item among the total number of responses per 100.
Depressive Symptoms | Immediately after the intervention
  Patient Health Questionnaire - 9. A self-applied questionnaire that identifies the presence of depressive symptomatology based on a Likert-type scale of 9 items. Based on the cut-off points, minimal (0-4), mild (5-9), moderate (10-14), moderate to severe (15-19) and severe (20-27) depression can be identified.
Anxiety symptoms | Immediately after the intervention
  General Anxiety Disorder - 7. A self-applied scale to identify generalized anxiety. It consists of a self-applied questionnaire of seven Likert-type questions. Based on the cut-off points, no anxiety (0-4), mild anxiety symptoms (5-9), moderate anxiety symptoms (10-14) and severe anxiety symptoms (15-21) can be identified.
Daily functionality | Immediately after the intervention
  The Activities of Daily Living Questionnaire. This instrument evaluates daily functioning by assessing basic and instrumental activities in six areas (self-care, home activities, work, recreation, money management, travel and communication, and information technology); it is usually useful for patients with mild cognitive or motor limitations. It allows to generate a percentage of functional impairment by adding the scores of each item among the total number of responses per 100.
Depressive Symptoms | Up to 12 weeks
  Patient Health Questionnaire - 9. A self-applied questionnaire that identifies the presence of depressive symptomatology based on a Likert-type scale of 9 items. Based on the cut-off points, minimal (0-4), mild (5-9), moderate (10-14), moderate to severe (15-19) and severe (20-27) depression can be identified.
Anxiety symptoms | Up to 12 weeks
  General Anxiety Disorder - 7. A self-applied scale to identify generalized anxiety. It consists of a self-applied questionnaire of seven Likert-type questions. Based on the cut-off points, no anxiety (0-4), mild anxiety symptoms (5-9), moderate anxiety symptoms (10-14) and severe anxiety symptoms (15-21) can be identified.
Daily functionality | Up to 12 weeks
  The Activities of Daily Living Questionnaire. This instrument evaluates daily functioning by assessing basic and instrumental activities in six areas (self-care, home activities, work, recreation, money management, travel and communication, and information technology); it is usually useful for patients with mild cognitive or motor limitations. It allows to generate a percentage of functional impairment by adding the scores of each item among the total number of responses per 100.

OTHER OUTCOMES:
Evaluation of the achievement of intervention objectives | Baseline
  Goal Assessment Scale. Mathematical technique that identifies the achievement of objectives in a rehabilitation program based on the perception of the patient and/or family member. Each objective is measured on a 5-point scale ranging from -2 to +2 (very little, little, expected level, more than expected, much more than expected).
Evaluation of the usability of the cognitive stimulation program | Immediately after the intervention
  System usability scale. A 5-level Likert-type scale (strongly disagree to strongly agree) that evaluates the opinion of the participants regarding the usability of digital systems. A maximum total score of 100 is obtained by averaging each response from all questionnaires.
Evaluation of the acceptability of the cognitive stimulation program | Immediately after the intervention
  In the last session of the intervention, a qualitative interview will be conducted with the participants. The interview will include questions associated with the relevance, usefulness, acceptability and satisfaction of the cognitive stimulation program.
Evaluation of the achievement of intervention objectives | Immediately after the intervention
  Goal Assessment Scale. Mathematical technique that identifies the achievement of objectives in a rehabilitation program based on the perception of the patient and/or family member. Each objective is measured on a 5-point scale ranging from -2 to +2 (very little, little, expected level, more than expected, much more than expected).

CONTACTS AND LOCATIONS:
Overall Officials: Natalia C Cortés, MD, Principal Investigator — Universidad Nacional Autonoma de Mexico; Ma Guillermina T Yáñez, PhD, Study Chair — Universidad Nacional Autonoma de Mexico; Dulce María Bélen C Prieto, PhD, Study Chair — Universidad Nacional Autonoma de Mexico; Edgar R Landa, PhD, Study Chair — Universidad Nacional Autonoma de Mexico; Juan C Castillo, PhD, Study Chair — National Polythecnic Institute
Locations (1):
- Condesa Iztapalapa Specialized Clinic, Mexico City, Iztapalapa, Mexico

IPD SHARING:
Plan to Share IPD: No
While the results of the present research will be shared in a scientific publication article, there is still no plan to make IPDs available due to the confidentiality that must be maintained when working with HIV+ populations and the ethical issues that remain during the research.

REFERENCES:
- [Background] Becker JT, Dew MA, Aizenstein HJ, Lopez OL, Morrow L, Saxton J, Tarraga L. A pilot study of the effects of internet-based cognitive stimulation on neuropsychological function in HIV disease. Disabil Rehabil. 2012;34(21):1848-52. doi: 10.3109/09638288.2012.667188. Epub 2012 Mar 30. PMID 22458375
- [Background] Bilder RM, Postal KS, Barisa M, Aase DM, Cullum CM, Gillaspy SR, Harder L, Kanter G, Lanca M, Lechuga DM, Morgan JM, Most R, Puente AE, Salinas CM, Woodhouse J. InterOrganizational practice committee recommendations/guidance for teleneuropsychology (TeleNP) in response to the COVID-19 pandemic. Clin Neuropsychol. 2020 Oct-Nov;34(7-8):1314-1334. doi: 10.1080/13854046.2020.1767214. Epub 2020 Jul 16. PMID 32673163
- [Background] Boivin MJ, Busman RA, Parikh SM, Bangirana P, Page CF, Opoka RO, Giordani B. A pilot study of the neuropsychological benefits of computerized cognitive rehabilitation in Ugandan children with HIV. Neuropsychology. 2010 Sep;24(5):667-73. doi: 10.1037/a0019312. PMID 20804255
- [Background] Vance DE, Fazeli PL, Ross LA, Wadley VG, Ball KK. Speed of processing training with middle-age and older adults with HIV: a pilot study. J Assoc Nurses AIDS Care. 2012 Nov-Dec;23(6):500-10. doi: 10.1016/j.jana.2012.01.005. Epub 2012 May 11. PMID 22579081
- [Background] Weber E, Blackstone K, Woods SP. Cognitive neurorehabilitation of HIV-associated neurocognitive disorders: a qualitative review and call to action. Neuropsychol Rev. 2013 Mar;23(1):81-98. doi: 10.1007/s11065-013-9225-6. Epub 2013 Feb 16. PMID 23417497
- [Background] Lancaster GA, Dodd S, Williamson PR. Design and analysis of pilot studies: recommendations for good practice. J Eval Clin Pract. 2004 May;10(2):307-12. doi: 10.1111/j..2002.384.doc.x. PMID 15189396
- [Background] Julious SA. Sample size of 12 per group rule of thumb for a pilot study. Pharmaceutical Statistics. 2005; 4: 287e91.
- [Background] Berryman A, Rasavage K, Politzer T, Gerber D. Oculomotor Treatment in Traumatic Brain Injury Rehabilitation: A Randomized Controlled Pilot Trial. Am J Occup Ther. 2020 Jan/Feb;74(1):7401185050p1-7401185050p7. doi: 10.5014/ajot.2020.026880. PMID 32078510
- [Background] Delaney MC. Caring for the caregivers: Evaluation of the effect of an eight-week pilot mindful self-compassion (MSC) training program on nurses' compassion fatigue and resilience. PLoS One. 2018 Nov 21;13(11):e0207261. doi: 10.1371/journal.pone.0207261. eCollection 2018. PMID 30462717
- See also: Joint United Nations Programme on HIV/AIDS (UNAIDS) (2018). Global AIDS update 2019. — https://www.unaids.org/sites/default/files/media_asset/UNAIDS_FactSheet_es.pdf
- See also: National Center for Prevention and Control of HIV and AIDS (CENSIDA) (2022). Epidemiological Surveillance of HIV/AIDS Cases in Mexico, Update for the 1st Quarter of 2022. — https://www.gob.mx/cms/uploads/attachment/file/750178/Informe_Hist_rico_VIH_DVEET_1er_TRIMESTRE_2022_Frev.pdf